CLINICAL TRIAL: NCT06632821
Title: The Relationship Between Health Literacy, Physical Activity, Back Pain and Posture Habits in University Students
Status: Not yet recruiting | Type: Observational
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Other Study IDs: health literacy
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: University Students
Keywords: university students; physical activity; back pain; posture habits
MeSH Terms: conditions — Motor Activity; Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University Students: Evaluation of university students' health literacy, physical activity, back pain and posture habits.
  Interventions: Other: No intervention will be used.

INTERVENTIONS:
Other: No intervention will be used. — University students' health literacy, physical activity, back pain and posture habits will be evaluated.

SUMMARY:
This study aims to investigate the relationship between health literacy, physical activity, back pain, and posture habits among university students. The Health Literacy Scale, the International Physical Activity Questionnaire, and the Posture Habits Questionnaire for Back Health in Daily Activities will be used to collect data from participants. Health literacy will be assessed in terms of individuals' ability to access, understand, and apply health-related information, while physical activity levels and posture habits will be examined for their influence on back pain. The findings are expected to shed light on the role of health literacy in promoting healthier physical activity and posture habits, providing insights for strategies to improve back health in this population.

ELIGIBILITY:
Inclusion Criteria:

* Being a university student

Exclusion Criteria:

* Having any diagnosed physical or psychological illness

Ages: 17 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: university students
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-21 (Estimated); Primary Completion 2024-12-09 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Health Literacy Scale | one month
  The Health Literacy Scale is comprised of 25 items, which are organised into four subscales. The scale comprises four subscales, namely access to information (items 1-5), understanding information (items 6-12), appraisal/evaluation (items 13-20) and application/use (items 21-25). The total score that can be obtained from the scale varies between 25 and 125 points. As the score obtained from the scale increases, the level of health literacy of the individual also increases.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | one month
  It is a short form consisting of 7 questions covering the last week in the assessment of physical activity level. The calculation of the total score of the short form includes the sum of the duration (minutes) and frequency (days) of walking, moderate intensity activity and intensity activity. The sitting score is calculated separately. The survey includes questions about PA performed for at least 10 minutes in the last week. A score is obtained as "MET-minutes/week" by multiplying minutes, days and MET values.
Posture Habits Questionnaire Related to Back Health in Daily Activities | one month
  The questionnaire was devised with the objective of evaluating the typical postural habits exhibited during the course of daily activities. The questionnaire comprises 31 questions. Four questions pertain to activities undertaken while standing, nine to activities performed while sitting, 13 to activities involving weight bearing, and five to activities carried out while lying down.